CLINICAL TRIAL: NCT01155271
Title: Comparison of 3 Exercise Training Modalities in Obese Patient With Sleep Apnea Syndrome Treated by Continue Positive Airway Pressure : a Randomized Controlled Study
Brief Title: OBese Patients With Obstructive Sleep Apnea Syndrome(OSAS) and EXercise Training
Acronym: OBEX1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AGIR à Dom (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGIR-03
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Sleep Apnea
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERGO (Active Comparator): General endurance training on cycloergometer
  Interventions: Other: Rehabilitation
- ERGONIV/ ERGOSPIRO (Active Comparator): General endurance training on cycloergometer using ventilatory assistance (ERGONIV) or additional respiratory muscle training (ERGOSPIRO)
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — 12 weeks : 3 sessions per week (2 supervised sessions and 1 session at home)
  1 technical visit and 1 nursing visit every two months at home for the CPAP

SUMMARY:
The study was designed to test the following hypotheses:

In obese patients with OSAS, the benefit of the combination of exercise training + continuous positive airway pressure (CPAP) will be higher than CPAP alone in term of functional capacity, metabolic, inflammatory, cardiovascular and sleep parameters and quality of life.

In obese patients with OSAS, the benefit of training using ventilatory assistance (NIV) during cycloergometer [cycloergometer with NIV] or respiratory muscles training (spirotiger) in addition to cycloergometer [cycloergometer + spirotiger] will be higher than cycloergometer training alone [cycloergometer] in term of functional and exercise capacities.

Dyspnea during walking test and respiratory muscle strength at baseline could influence the response to combined exercise training such as [cycloergometer + NIV] or [cycloergometer + spirotiger]

DETAILED DESCRIPTION:
Background: Obesity and sleep apnea syndrome lead to metabolic troubles and increasing cardiovascular risk. Furthermore, both diseases are associated with reduced exercise tolerance. We hypothesized that exercise training could be complementary to nocturnal ventilatory treatment in restoring metabolic disturbances, exercise tolerance and sleep parameters in obese patients with SAS.

Objective: To evaluate the effect of training on exercise tolerance (walking distance and dyspnea during walk)(main objective), systemic inflammation, vascular endothelial function, insulin resistance, quality of sleep and quality of life in obese patients treated by CPAP for OSAS (secondary objectives)

Methods: We proposed to conduct a controlled, randomized clinical trial comparing the efficacy of 3 different modalities of training in obese patients with SAS. After a 6-week control pre-inclusion period, patients are included in either [cycloergometer] vs. [cycloergometer with ventilatory assistance] vs. [cycloergometer + respiratory muscle exercises]. Before and after the control period, and both immediately and 9 month after training, patients perform walking test, maximal incremental test on cycloergometer, blood sampling and cardiovascular function, body composition, muscle function, quality of sleep and quality of life assessments as well as spontaneous physical activity measurement. During the 5 years following inclusion in the training program, the number of cardiovascular event is recorded every year.

An interim analysis will be carried out when 30 will have completed the third evaluation session (after the training program). The Peto's method will be used to correct the p-values.

ELIGIBILITY:
Inclusion Criteria:

* OSAS (AHI > 30 before CPAP treatment)
* > 4h/d CPAP treatment adherence
* Obese patients with 35 < BMI < 45 kg/m2
* Patients who give written consent
* Patients who subscribed social insurance

Exclusion Criteria:

* Cardiovascular or respiratory failure discovered at the moment of the inclusion in the study
* Contraindication to exercise
* Pregnant or breast-feed woman
* Patients under guardianship
* Imprisoned patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in exercise tolerance during walking test | After control period (6th wk) vs. after training period (18th wk)
  * walking distance
  * dyspnea score

SECONDARY OUTCOMES:
Changes in Aerobic capacity | After control period (6th wk) vs. after training period (18th and 52th wks)
  Maximal oxygen consumption
Changes in cardiovascular and metabolic function | After control period (6th wk) vs. after training period (18th and 52th wks)
  Pulse wave velocity, peripheral arterial tone, BP, inflammatory and metabolic plasmatic markers
Changes in sleep parameters and Quality Of life | After control period (6th wk) vs. after training period (18th and 52th wks)
  Nocturnal oxygen saturation, CPAP data, Epworth questionnaire, Short Form (36) Health Survey questionnaire
Number of cardiovascular events per year | Every year from the 1st to the 5th year
  Questionnaire sent to the patient by mail
Changes in body composition | After control period (6th wk) vs. after training period (18th and 52th wks)
  Fat mass and fat-mass index Fat-free mass and fat-free mass index assessed by impedancemetry measurements
Change in physical activity and sleep duration | After control period (6th wk) vs. after training period (18th and 52th wks)
  Number of hour per day of physical activity at 1, 2, 3 or 4 Metabolic Equivalents (METS); Number of steps per day; Sleep to lying position duration ratio
Change in exercise tolerance during walking test | After control period (6th wk) vs. after trainng (52th wk)
  * isotime dyspnea
  * isotime oxygen saturation
Change in physiological variables during the control period | Before (1st) vs. after control period (6th wk)
  * functional and exercise parameters
  * cardiovascular parameters
  * metabolic parameters
  * sleep and quality of life parameters (Short Form (36) Health Survey)
  * physical activity
Baseline characteristics | Before control period (1st week) or after the control period (6th week)
  * functional and exercise parameters
  * cardiovascular parameters
  * metabolic parameters
  * sleep and quality of life parameters (Short Form (36) Health Survey)
  * physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pepin, MD, PhD, Principal Investigator — Laboratoire EFCR, CHU de Grenoble, 38043, Grenoble, France
Locations (2):
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec, Canada
- Hopital Universitaire de Grenoble, Grenoble, France

REFERENCES:
- [Derived] Vivodtzev I, Tamisier R, Croteau M, Borel JC, Grangier A, Wuyam B, Levy P, Minville C, Series F, Maltais F, Pepin JL. Ventilatory support or respiratory muscle training as adjuncts to exercise in obese CPAP-treated patients with obstructive sleep apnoea: a randomised controlled trial. Thorax. 2018 Feb 20:thoraxjnl-2017-211152. doi: 10.1136/thoraxjnl-2017-211152. Online ahead of print. PMID 29463621